CLINICAL TRIAL: NCT01170299
Title: A Randomized Controlled Trial to Investigate the Role of Low or High 'Fibre' Diets in Patients Undergoing Pelvic Radiotherapy - The Fibre Study
Brief Title: Low-Fiber Diet or High-Fiber Diet in Preventing Bowel Side Effects in Patients Undergoing Radiation Therapy for Gynecological Cancer, Bladder Cancer, Colorectal Cancer, or Anal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: RM-FIBRE-STUDY; CDR0000681693 (Registry Identifier: PDQ (Physician Data Query)); RM-CCR-3142; EU-21053
Record Dates: First submitted 2010-07-24; First posted 2010-07-27 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2010-07

CONDITIONS: Anal Cancer; Bladder Cancer; Cervical Cancer; Colorectal Cancer; Fallopian Tube Cancer; Gastrointestinal Complications; Ovarian Cancer; Radiation Toxicity; Sarcoma
Keywords: radiation toxicity; gastrointestinal complications; cervical cancer; fallopian tube cancer; ovarian epithelial cancer; ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; uterine sarcoma; bladder cancer; colon cancer; rectal cancer; anal cancer
MeSH Terms: conditions — Anus Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Radiation Injuries; Sarcoma; Carcinoma, Ovarian Epithelial; Colonic Neoplasms; Rectal Neoplasms | interventions — Diet Therapy; Serotonin Plasma Membrane Transport Proteins

INTERVENTIONS:
Dietary Supplement: dietary intervention
Other: laboratory biomarker analysis
Procedure: gastrointestinal complications management/prevention
Procedure: management of therapy complications
Radiation: selective external radiation therapy

SUMMARY:
RATIONALE: Fiber may lessen bowel side effects caused by radiation therapy. It is not yet known whether a high-fiber diet is more effective than a low-fiber diet in preventing bowel side effects caused by radiation therapy.

PURPOSE: This randomized clinical trial is studying a high-fiber diet to see how well it works compared with a low-fiber diet in preventing bowel side effects in patients undergoing radiation therapy for gynecological cancer, bladder cancer, colorectal cancer, or anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of a high- vs low-fiber intervention in preventing bowel toxicity in patients receiving radical pelvic radiotherapy treatment for gynecological, urological (bladder), colorectal, or anal malignancy.
* To compare whether a high- or low-fiber intervention has any beneficial effect over no intervention (i.e., ad-libitum fiber consumption).
* To examine the effect of a low- or high-fiber diet on gastrointestinal symptoms, measured using the IBDQ-B and Bristol Stool Chart, in patients receiving radical radiotherapy for pelvic malignancies.
* To minimize any potential risk associated with change in fiber intake by using a controlled and gradual dietary-based intervention combined with dietetic advice.

Secondary

* To examine the relationship between volume of irradiated bowel and onset of gastrointestinal symptoms as measured by the Bristol Stool Chart.
* To measure percentage compliance with fiber prescription through validated dietetic techniques including the 7-day Food Diary using household measures and the 24-hour recall.

OUTLINE: Patients are stratified according to disease (gynecological vs gastrointestinal) and concomitant therapy (received vs not received). Patients are randomized to 1 of 3 treatment arms.

* Arm I (low-fiber diet): Patients are assessed by a qualified dietitian, receive written guidance, and are counseled as to how best to meet their study fiber prescription of a low-fiber diet, comprising 'not more than' 10 g of fiber per day for up to 7 weeks.
* Arm II (high-fiber diet): Patients are assessed by a qualified dietitian, receive written guidance, and are counseled as to how best to meet their study fiber prescription of a high-fiber diet, comprising a target of between 18 and 22 g of fiber per day for up to 7 weeks.
* Arm III (no intervention): Patients receive advice designed to ensure they maintain their normal habitual diet for up to 7 weeks.

All patients undergo radiotherapy once daily comprising approximately 25 (or more) fractions in total to be delivered for 5-7 weeks in the absence of unacceptable toxicity.

All patients are asked to complete two 7-day Food Diaries at baseline and end of radiotherapy treatment. All patients keep a daily record of stool characteristics and frequency using the Bristol Stool Chart. Patients also complete a short 1-page weekly-cost questionnaire to assess the economic impact of symptom management. Patients in arms I and II complete several additional questions regarding the costs (if any) of adhering to their fiber prescription and the palatability of the diet.

Blood and stool samples may be collected at baseline and during study therapy for biomarker analysis.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gynecological, urological (bladder), colorectal, or anal malignant cancer
* Scheduled to undergo a course of radical or adjuvant pelvic radiotherapy (≥ 45 Gy)

  * Radiotherapy regimen will be delivered in daily fractions comprising approximately ≥ 25 fractions over 5-7 weeks

PATIENT CHARACTERISTICS:

* No prior prescribed low-residue diet for a clear medical reason
* No established wheat intolerance or celiac disease
* No concurrent condition precluding oral nutritional intake

PRIOR CONCURRENT THERAPY:

* No gastrointestinal stent
* No jejunostomy, ileostomy, or colostomy
* No concurrent participation in a study with toxicity as an endpoint

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in IBDQ-B (Inflammatory Bowel Disease Questionnaire - Bowel Subset) score between baseline (i.e., Day 1 of radiotherapy treatment) and the nadir score during treatment

SECONDARY OUTCOMES:
Incidence of toxicity, defined using the Bristol Stool Chart
Costs for symptom management

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Blake, MD, Study Chair — Royal Marsden NHS Foundation Trust; Jervoise Andreyev, MD — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom